CLINICAL TRIAL: NCT05135117
Title: Impact of Neck Cooling Collar on Exercise Performance in the Heat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: NeuroRescue Inc. (Unknown)
Responsible Party: Principal Investigator, Douglas J Casa, Principal Investigaator, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H21-0053
Record Dates: First submitted 2021-09-26; First posted 2021-11-26 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Passive rest - no intervention provided
- Ice towel cooling (Active Comparator): About 6-12 cooling periods of ice towel lasting between 5-20 minutes will be done and equally distributed throughout the respective trials. Towels dipped in ice water will be placed on subjects necks during this time.
  Interventions: Other: Ice Towel
- NeuroRescue Neck Cooling Collar (Experimental): About 6-12 cooling periods of neck cooling with the NeuroRescue collar lasting between 5-20 minutes will be done and equally distributed throughout the respective trials.
  Interventions: Other: NeuroRescue Cooling Collar

INTERVENTIONS:
Other: NeuroRescue Cooling Collar — Between bouts of exercise subjects will be provided cooling on the neck with the NeuroRescue Collar. The custom sized cooling collar has ice water (which is kept around 2 degrees celsius) that is circulated through a neoprene sleeve that is attached to their neck for the cooling period.
  Arms: NeuroRescue Neck Cooling Collar
Other: Ice Towel — Between bouts of exercise subjects will be provided cooling on the neck with a towel. The towel will be kept in ice water (which is kept around 2 degrees celsius) and placed around the neck of the individual during the cooling intervention period.
  Arms: Ice towel cooling

SUMMARY:
During exercise in the heat, the thermoregulatory system impacts performance in an athletic population. Increased in core body temperature could lead to development of heat-related illnesses and impair physical performance. To facilitate heat loss and optimize performance during exercise in the heat, various cooling strategies, including cold water immersion and wearable cooling devices have been previously explored. Although whole body cooling by cold water immersion is considered to be the most effective way to reduce core body temperature, this cooling method would not be feasible for athletes during practice or competition. Therefore, previous studies strongly recommended neck cooling during exercise because of the rate of heat dissipation through the large blood vessel and accessibility compared to other body part. Furthermore, multiple studies reported that the neck cooling could improve aerobic performance (i.e. running distance and time). In addition to physiological changes, human prefer to be cool in the neck region as well as the face in hot environment. Thus, local cooling of the neck is efficient way to reduce thermal discomfort during heat exposure. The novel neck cooling collar device (NeuroRescue Inc., Lafayette, LA) used in the current study may be able to produce powerful effect of conductive cooling, which result in improving performance and also reduce thermal discomfort during exercise in the heat.

While this neck cooling collar would assist athletes in improving sports safety and performance by decreasing skin temperature around the neck, the effectiveness of this neck cooling collar on core temperature was not examined at this point. Moreover, other physiological and perceptual changes are important to assess along with changes in core body temperature. Therefore, this study aims to examine how internal body temperature, heart rate, perceptual measures, and athletic performance are affected by the novel neck cooling collar during exercise in the heat.

ELIGIBILITY:
Inclusion Criteria:

1. Physically active (at least 30 minutes of exercise 3-5 days per week) male
2. been cleared by the medical monitor for this study
3. Have a VO2max >45ml/kg/min

Exclusion Criteria:

1. Have a current musculoskeletal injury that would limit their physical activity or preclude the participant from walking, jogging, running, sprinting, or cutting.
2. Chronic health problems that affect your ability to thermoregulate (disorders affecting the liver, kidneys or the ability to sweat normally)
3. Fever or current illness at the time of testing
4. History of cardiovascular, metabolic, or respiratory disease
5. A family member died for no apparent reason, had a heart attack, died from heart problems, or sudden death before the age of 50
6. Current musculoskeletal injury that limits their physical activity
7. Currently taking a medication that is known to influence body temperature (amphetamines, antihypertensives, anticholinergics, acetaminophen, diuretics, NSAIDs, aspirin)
8. Are a female. Due to the internal body temperature gradient that accompanies the menstrual cycle, inclusion of females may not provide the most controlled internal body temperature data for this study.
9. Have a history of heat related illness
10. Throat or gastroesophageal diseases including gastroesophageal reflux disease (aka, GERD) or difficulty swallowing
11. Have any allergies or adverse reactions to the cold (e.g. Cold Urticaria, Raynauds Phenomenon/Disease, or cryoglobulinaemia)
12. Any COVID-19 related symptoms including fever, cough, shortness of breath or difficulty breathing, gastrointestinal discomfort (nausea, vomiting, and/or diarrhea), repeated shaking with chills, muscle pain (unrelated to exercise), headache, sore throat, new loss of taste or smell, congestion or runny nose.
13. Participant with clinical diagnosis of COVID-19 infection or positive result on a COVID-19 test due to concern about cardiac complications.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Esophageal Temperature Change | Up to 4 weeks
  Esophageal Temperature Change

SECONDARY OUTCOMES:
Rectal Temperature Change | Up to 4 weeks
  Rectal Temperature Change
Heart Rate Change | Up to 4 weeks
  Heart rate as beats per minute Change
Performance Test Change | Up to 4 weeks
  Reaction Time Test
Performance Test Change | Up to 4 weeks
  Broad jump
Performance Test Change | Up to 4 weeks
  Agility test
Performance Test Change | Up to 4 weeks
  15-min time trial
Perceptual Scale Change | Up to 4 weeks
  Rating of Perceived Exertion (6-20, lower exertion indicated by lower number)
Perceptual Scale Change | Up to 4 weeks
  Thermal Sensation Scale (0-8, lower number indicates cooler, higher number indicates hotter sensations)
Perceptual Scale Change | Up to 4 weeks
  Thirst Scale (1-9, 1 indicates not thirst, 9 indicates very very thirsty)
Perceptual Scale Change | Up to 4 weeks
  Fatigue Scale (0-10, 0 indicates no fatigue, 10 indicates extreme fatigue)
Perceptual Scale Change | Up to 4 weeks
  Environmental Symptoms questionnaire (0-70, 0 indicates no heat stress)
Perceptual Scale Change | Up to 4 weeks
  Profile of mood states (0-260, 0 indicates lower mood disturbance)
Cognitive Functioning Change - Automated Neuropsychological Assessment Metrics (ANAM) Test System | Up to 4 weeks
  Go/No Go (0-infinity, lower number indicates faster and more accurate response)
Cognitive Functioning Change- Automated Neuropsychological Assessment Metrics (ANAM) Test System | Up to 4 weeks
  Spatial Processing (0-infinity, lower number indicates faster and more accurate response)
Cognitive Functioning Change- Automated Neuropsychological Assessment Metrics (ANAM) Test System | Up to 4 weeks
  Stroop (0-infinity, lower number indicates faster and more accurate response)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No